CLINICAL TRIAL: NCT01361581
Title: Metabolic Aspects of Citrate Anticoagulation in Renal Replacement Therapy
Acronym: Citrate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: Martin Balik, A/Prof., MD, PhD, EDIC, 1st Medical Faculty, Charles University, Prague
Other Study IDs: NS/10014-4
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Acute Renal Failure; Critical Illness
Keywords: Acute renal failure; Anticoagulation; Citrate; Haemodiafiltration; Haemofiltration; Renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ACD (acid-citrate-dextrose)
- 4% trisodium citrate
- unfractionated heparin (UFH)

SUMMARY:
Citrate anticoagulation is associated with metabolic side effects which are linked to a portion of citrate reaching systemic circulation. Data on significance of systemic gain of citrate and its relationship to method configuration are missing. Patient might also receive certain dose of lactate as a buffer and a dose of glucose if acid-citrate-dextrose solution is used. The authors test variable methods of indirect estimate of systemic dose of citrate which would allow to quantify the metabolic input without mostly unavailable measurements of citrate levels.

ELIGIBILITY:
Inclusion Criteria:

* Acute renal failure on continuous renal replacement therapy for more than 24 hours (CVVH or CVVHDF).

Exclusion Criteria:

* Absence of consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: critically ill intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-01

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anaesthesia and Intensive Care, General University Hospital, 1st Medical Faculty, Charles University, Prague, Czechia

REFERENCES:
- [Derived] Zakharchenko M, Los F, Brodska H, Balik M. The Effects of High Level Magnesium Dialysis/Substitution Fluid on Magnesium Homeostasis under Regional Citrate Anticoagulation in Critically Ill. PLoS One. 2016 Jul 8;11(7):e0158179. doi: 10.1371/journal.pone.0158179. eCollection 2016. PMID 27391902
- [Derived] Balik M, Zakharchenko M, Leden P, Otahal M, Hruby J, Polak F, Rusinova K, Stach Z, Tokarik M, Vavrova J, Jabor A, Oudemans-van Straaten HM. Bioenergetic gain of citrate anticoagulated continuous hemodiafiltration--a comparison between 2 citrate modalities and unfractionated heparin. J Crit Care. 2013 Feb;28(1):87-95. doi: 10.1016/j.jcrc.2012.06.003. Epub 2012 Aug 27. PMID 22951019